CLINICAL TRIAL: NCT05243433
Title: Maestro LIFT-OFF: A Feasibility, Prospective, Single Center, Single-arm Study of the Maestro Surgical Assistance Device in Abdominal Laparoscopic Surgery
Brief Title: Maestro LIFT-OFF: Surgical Assistance Device in Abdominal Laparoscopic Surgery
Acronym: Maestro
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Moon Surgical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Maestro LIFT-OFF
Record Dates: First submitted 2022-01-12; First posted 2022-02-17 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Surgery
Keywords: abdominal laparoscopic surgery; laparoscopic cholecystectomy; laparoscopic hernia repair; laparoscopic appendectomy; laparoscopic bariatric surgery; laparoscopic colectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Procedure using the Maestro Platform (Experimental): Study participants will be adults aged ≥ 18 to ≤ 75 years scheduled for a non-emergent laparoscopic cholecystectomy, laparoscopic hernia repair, laparoscopic appendectomy, laparoscopic bariatric surgery (gastric sleeve or gastric bypass), or laparoscopic colectomy.
  Interventions: Device: Laparoscopic surgery using the Maestro Platform

INTERVENTIONS:
Device: Laparoscopic surgery using the Maestro Platform — Laparoscopic cholecystectomy, laparoscopic hernia repair, laparoscopic appendectomy, laparoscopic bariatric surgery (gastric sleeve or gastric bypass), or laparoscopic colectomy performed using the Maestro Platform.

SUMMARY:
The objective of the study is to provide evidence for the safety and effectiveness of the Maestro Platform for surgical assistance in abdominal laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 18 to ≤ 75 years
* Scheduled for one of the following non-emergent laparoscopic procedure: cholecystectomy, hernia repair, appendectomy, bariatric surgery (gastric sleeve or gastric bypass), or colectomy.
* Willing to comply with protocol-specified follow-up evaluation
* Signed informed consent

Exclusion Criteria:

* Advanced refusal of blood transfusion, if necessary;
* Active systemic or cutaneous infection or inflammation;
* Pre-existing immunodeficiency disorder and/or chronic use of systemic steroids;
* Uncontrolled diabetes mellitus;
* Known, significant history of bleeding diathesis, or coagulopathy, or Von Willebrand's disease or current platelet count < 100,000 cells/mm3, or baseline INR ≥1.8, or fibrinogen level less than 150 mg/dl (if received a fibrinolytic agent within prior 24 hours);
* Severe co-existing morbidities having a life expectancy of less than 30 days;
* Currently participating in another investigational drug or device study that clinically interferes with the endpoints of this study;
* Significant anemia with a hemoglobin level less than 10 g/dL or a hematocrit less than 30%;
* Renal insufficiency (serum creatinine of > 2.5 mg/dl);
* Females who are pregnant, planning to become pregnant within three months of the procedure, or lactating;
* Extreme morbid obesity (BMI greater than 45 kg/m2);
* Patients presenting with ascites;
* Patients presenting for emergency surgery;
* Previous surgery in the same anatomical location;
* Lack of capacity to give informed consent (individuals deprived of their liberty subject to a legal protection measure or who are unable to express their consent, individuals under guardianship or curatorship)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2023-04-05 (Actual); Study Completion 2023-05-05 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) in terms of type (device/procedure related), seriousness, level of severity. Rate of occurence of intra-procedural and post-procedural adverse events, and device related complications | 30 days
Completion of the procedure using the Maestro Platform without conversion to a manual minimally invasive or open surgical procedure specifically due to a device failure or malfunction | During procedure

OTHER OUTCOMES:
Procedure-specific complications | During procedure
Procedure duration | During procedure
Recovery time | 30 days
Post-operative pain (Visual analogue scale 0 - no pain to 10 - worst pain possible) | 1 day after procedure
Number of rehospitalization per patient within 30 days | 30 days
Number of repeat surgery or reintervention per patient within 30 days | 30 days
Surgeon comfort evaluated on 1-10 scale at the end of the procedure (1-not comfortable, 10-very comfortable) | During procedure
Surgeon satisfaction with the level of assistance provided by the Maestro platform, on 1-10 scale at the end of the procedure (1-assistance much worse than a human assistant, 5-equivalent to human assistant, 10-much better than human assistant) | During procedure
Study device usability on 1-10 scale at the end of the procedure (1-very hard to use, 5-not difficult but not easy, 10-very easy to use) | During procedure

CONTACTS AND LOCATIONS:
Overall Officials: Guy-Bernard CADIERE, Pr, Principal Investigator — CHU Saint-Pierre, Brussels, Belgique
Locations (1):
- CHU St Pierre, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided